CLINICAL TRIAL: NCT02264431
Title: Determinants of Nocturnal Respiratory Disorders of Obese Patients Referred to in a Specialized Center.
Brief Title: Severe Obesity Outcome Network Cohort (SOON)
Acronym: SOON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Act For Chronic Diseases (Other); HP2 laboratory INSERM U1042 (Unknown); University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 1327; 2013-A01097-38 (Registry Identifier: n°ID RCB)
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Obstructive Sleep Apnea; Sleep
Keywords: Obesity; Obstructive Sleep Apnea; Sleep Habits; Bariatric Surgery; Cohort
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum bank, gene bank, tissue bank (subcutaneous fat, visceral fat)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to identify the determinant of sleep characteristics of obese patients attempting a tertiary clinical center for obesity management, including bariatric surgery.

More accurately the questions addressed are:

* What are the determinants of the sleep habits (sleep duration, chronotype) and of their evolution
* What are the determinants of sleep breathing disorders (sleep apnea, obesity hypoventilation syndrome) and of their evolution

DETAILED DESCRIPTION:
Adult obese patients, attempting a tertiary medical center for the management of their obesity, are asked to participate in a cohort study. Data issued from routine clinical practice are collected.

Medical history and actual medical condition:

* Type 2 or type 1 diabetes
* Dyslipidemia
* Hypertension
* Cardiovascular diseases
* Steatohepatitis/cirrhosis
* Gastric disorders
* Nutritional deficiency
* Obstructive sleep apnea/Obesity hypoventilation syndrome

All patients who do not have a previously known sleep apnea syndrome are evaluated by nocturnal polygraphy.

Lifestyle and sleep habits, as well as social and economic characteristics, are assessed by questionnaires.

Patients are asked to provide blood sample to constituate a serum bank and gene bank.

Patients are asked, if undergoing bariatric surgery, to provide subcutaneous and visceral fat.

When patients benefit from bariatric surgery, follow-up data are collected at 3 months, 6 months, 12 months after bariatric surgery and yearly after that for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Class II or class III obesity (BMI ≥ 35 kg/m²). Only patients undergoing surgery to realize a second surgical line of management of their obesity may have a lower BMI, if the surgical recovery is motivated by a technical defect of the first assembly.

Exclusion Criteria:

* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with class II or class III obesity (Body mass index ≥ 35kg/m²)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Sleep breathing disorders | 5 years
  Evolution of sleep breathing disorders during obesity management, especially after bariatric surgery

SECONDARY OUTCOMES:
Sleep habits | 5 years
  Evolution of sleep habits during obesity care, especially after bariatric surgery

OTHER OUTCOMES:
Metabolic diseases | 5 years
  Evolution of metabolic diseases during obesity care, especially after bariatric surgery
Other respiratory diseases | 5 years
  Evolution of other respiratory diseases during obesity care, especially after bariatric surgery
Complications of bariatric surgery | 5 years
  Recording of complications after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Borel, Pr MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borel AL, Van Ngo TH, Coumes S, Pepin JL, Abba J, Tamisier R, Tonetti G, Suzeau P, Reche F, Bailly S. Cluster analysis in subjects living with obesity and association with bariatric surgery outcomes: The severe obesity outcome network cohort. Clin Nutr. 2025 Nov;54:210-219. doi: 10.1016/j.clnu.2025.09.022. Epub 2025 Oct 4. PMID 41092584
- [Derived] Guggino J, Coumes S, Wion N, Reche F, Arvieux C, Borel AL. Effectiveness and Safety of Bariatric Surgery in Patients with End-Stage Chronic Kidney Disease or Kidney Transplant. Obesity (Silver Spring). 2020 Dec;28(12):2290-2304. doi: 10.1002/oby.23001. PMID 33230959